CLINICAL TRIAL: NCT06297200
Title: Investigations of Low-Intensity Focused Ultrasound Towards Treatment for the Complex Patient
Brief Title: Low-Intensity Focused Ultrasound and the Complex Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Salem VA Medical Center (Unknown); Washington DC VA Medical Center (Unknown)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-050
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Chronic Pain; Anxiety Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Masking Description: Sham trials will be utilized within subject. All subjects will receive sham and ultrasound conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Pain, Craving, and Anxiety measures (Experimental): Multi visit - LIFU/Sham. Participants will complete pain, craving, and anxiety measures pre and post intervention.
  Interventions: Device: Low-Intensity Focused Ultrasound; Device: Low-Intensity Focused Ultrasound - sham

INTERVENTIONS:
Device: Low-Intensity Focused Ultrasound — A noninvasive brain stimulation device using low-intensity focused ultrasound (LIFU) - ultrasound will be used to test whether noninvasive brain stimulation can effect pain, craving, and anxiety.
Device: Low-Intensity Focused Ultrasound - sham — A sham condition that will mimic the application of LIFU without actually administering any ultrasound to the brain.

SUMMARY:
Studying the effects of Low Intensity Focused Ultrasound (LIFU) on measures of pain, craving, and anxiety in a complex patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-65 years
2. Current diagnosis of Chronic Back Pain as defined by pain duration of at least three months, with back pain being an ongoing problem for at least half the days of the last six months.
3. Have evidence of central sensitization (CS) as measured by the Widespread Pain/Symptom Severity Index (WPSSI) with a score of Widespread Pain Index (WPI) ≥ 7 and Symptom Severity (SS) ≥ 5 or WPI = 3-6 and SS ≥ 9.
4. Meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for current opiate use disorder as diagnosed by the Structured Clinical Interview for DSM-5.
5. Be in treatment for opioid use disorder (OUD) including buprenorphine or methadone.
6. Meet the DSM-5 criteria for a current anxiety disorder: generalized anxiety disorder, post-traumatic stress disorder or social anxiety disorder as diagnosed by the Structured Clinical Interview for DSM-5.

Exclusion Criteria:

1. Evidence of neuropathic pain
2. Previous spine surgery
3. Current substance use disorder other than OUD or tobacco use disorder
4. Current DSM-5 diagnosis of schizophrenia or schizo-affective disorder
5. Chronic Pain Conditions other than chronic back pain
6. Daily opiate use other than buprenorphine/methadone for OUD/pain control
7. Pregnant or breastfeeding
8. History of head injury, seizures, neurologic disorders including cerebrovascular disease, stroke, brain surgery, brain tumor, multiple sclerosis, or neurodegenerative diseases
9. History of metastasizing cancers, inflammatory disorder (rheumatoid arthritis, polymyalgia rheumatica, scleroderma, lupus or polymyositis), unintended weight loss of 20 pounds or more in the last year, or cauda equina syndrome
10. Ferromagnetic implants or other contraindications for magnetic resonance imaging (MRI)
11. Evidence of arteriovenous malformation, aneurysm, infarct, meningioma, parenchymal brain tumor or evidence of neurodegenerative processes and/or white matter lesions greater than that expected for age as determined by the study neuroradiologist
12. Unstable medical conditions such as congestive heart failure, unstable angina, poorly controlled arrhythmia active system infection end stage renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events via a neurological examination | Assessed per participant, over the course of participation - an average of 4 weeks
  Any abnormal finding from the neurological exam will be recorded as an adverse event (AE) and tabulated with the side effects and tolerability data.
Incidence of Treatment-Emergent Adverse Events via a side effects questionnaire | Assessed per participant, over the course of participation - an average of 4 weeks
  Side effects and reported severity will be tabulated and summarized on a 5 point likert scale.
Changes in Heart Rate (HR) | Assessed per participant, over the course of participation - an average of 4 weeks
  changes in HR compared pre/post LIFU and at follow up
Changes in Respiration Rate (RR) | Assessed per participant, over the course of participation - an average of 4 weeks
  changes in RR compared pre/post LIFU and at follow up
Changes in mood via visual analog mood scale (VAMS) such as the wong-baker face scale. | Assessed per participant, over the course of participation - an average of 4 weeks
  changes in mood scale compared pre/post LIFU and at follow up
Changes in Blood Pressure (BP) | Assessed per participant, over the course of participation - an average of 4 weeks
  changes in BP (systolic and diastolic) compared pre/post LIFU and at follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No